CLINICAL TRIAL: NCT02571101
Title: A Prospective, Randomized, Double-blinded, Active-control, 3-Treatment Arm, Parallel, Multi-center, Phase 2 Trial to Evaluate Safety and Efficacy With CDFR0812-15/25mg and CDFR0812-15/50mg Compared to Clomipramine HCl 15mg in Male Patients Diagnosed With Premature Ejaculation
Brief Title: A Phase 2 Study of On-demand Therapy With Clomipramine and Sildenafil Combination in Premature Ejaculation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CTC Bio, Inc. (Industry)
Collaborators: Symyoo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTC-PED-CDFR0812_P2
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Premature Ejaculation
Keywords: Clomipramine; Premature ejaculation; CDFR0812; Sildenafil
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test 1 (Experimental): Test 1 subjects will take one tablet of CDFR0812-15/25mg and another tablet of Condencia-Placebo before sexual intercourse in on-demand for 8 weeks.
  Interventions: Drug: CDFR0812-15/25mg; Drug: Condencia-Placebo
- Test 2 (Experimental): Test 2 subjects will take one tablet of CDFR0812-15/50mg and another tablet of Condencia-Placebo before sexual intercourse in on-demand for 8 weeks.
  Interventions: Drug: CDFR0812-15/50mg; Drug: Condencia-Placebo
- Comparator (Placebo Comparator): Comparator subjects will take one tablet of Condencia and another tablet of CDFR0812-Placebo before sexual intercourse in on-demand for 8 weeks.
  Interventions: Drug: Condencia; Drug: CDFR0812-Placebo

INTERVENTIONS:
Drug: CDFR0812-15/25mg — Contains chlomipramine HCl 15mg and sildenafil citrate 25mg.
  Arms: Test 1
Drug: CDFR0812-15/50mg — Contains chlomipramine HCl 15mg and sildenafil citrate 50mg.
  Arms: Test 2
Drug: Condencia — Contains chlomipramine HCl 15mg.
  Arms: Comparator
Drug: CDFR0812-Placebo — Placebo tablet of CDFR0812.
  Arms: Comparator
Drug: Condencia-Placebo — Placebo tablet of Condencia
  Arms: Test 1; Test 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of on-demand therapy with CDFR0812-15/25mg and CDFR0812-15/50mg compared to on-demand therapy with single-drug administration of Clomipramine HCl 15mg in Korean Male Patients Diagnosed with Premature Ejaculation

DETAILED DESCRIPTION:
Clomipramine is a dibenzazepine-derivative tricyclic antidepressant (TCA) and is a potent inhibitor of serotonin and norepinephrine reuptake. Clomipramine may be used in a variety of indications. Condencia Tab contains low dose of 15mg of clomipramine HCl as an active ingredient, which is newly approved to market for the treatment of premature ejaculation. This study is a prospective, randomized, double-blinded, active-control, 3-treatment arm, parallel, multi-center clinical trial. Approximately a total of 297 male patients diagnosed with premature ejaculation will be enrolled and randomized into 3 groups (99 subjects per a group).

The efficacy of oral administration of Clomipramine HCl will be investigated closely compared to the effects after oral administration of CDFR0812-15/25mg and CDFR0812-15/50mg.

The secondary object is to investigate general safety of oral administration of CDFR0812-15/25mg and CDFR0812-15/50mg.

ELIGIBILITY:
Inclusion Criteria:

* Korean male aged between 19 and 65
* Both patient and his partner given their informed and written consents
* Patient who has persisted for at least 6 months and is willing to retain the relationship during this study
* Patient diagnosed with premature ejaculation according to DSM-V
* Patient whose score in PEDT (Korean version) is 11 and more
* Patient who are willing to try 4 and more intercourse attempts for Run-in period and he has experienced 75%-100% of the IELT within one minute or less of vaginal penetration
* Patient whose personal distress in PEP is 'moderate' and over.
* Patient who is willing to participate in the study by the end and are cooperative (trying 4 and more intercourse attempts between each visit and able to postpone scheduled elective surgery)
* Patient who is willing to complete a patient diary and questionnaires

Exclusion Criteria:

* Patient who has a medical history including neurological disorders, infectious diseases, damage, surgery or medication history and that is judged to be related to premature ejaculation
* Patient who has participated into other trials within 90 days before this study
* Patient who is in a unstable medical condition or has alcohol/drug abuse in recent 6 months
* Patient whose female partner is less interested in sexual intercourse or has a sexual disorder
* Patient whose female partner is pregnant
* Patient whose female partner of childbearing age is not willing to use proper birth control
* Patient whose IIEF-EF score is 25 and less
* Medical history of convulsive diseases, mental diseases, E.C.T (Electroconvulsive shock Treatment), glaucoma
* Patient who has taken concomitantly prohibited medicines before the study and who is not willing to stop the medications for appropriate wash-out period

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The fold change of IELT | From 4 weeks to 8 weeks after dosing
  IELT(Intravaginal Ejaculation Latency Time), which is to be reported through patient diary

SECONDARY OUTCOMES:
The % change of IELT | From 4 weeks to 8 weeks after dosing
  IELT(Intravaginal Ejaculation Latency Time), which is to be reported through patient diary
The mean change of IELT | From 4 weeks to 8 weeks after dosing
  IELT(Intravaginal Ejaculation Latency Time), which is to be reported through patient diary
The response rate | At 8 weeks after dosing
  PEP (Premature Ejaculation Profile) questionnaire
Global impression reported by patient | At 8 weeks after dosing
  PGIG (Patient Global Impression of Change in Premature Ejaculation)
Administration time of study drug | for 8 weeks
  The time when a patient takes study drug before sexual attempt
Number of patients with adverse events | for 8 weeks
  It will be assessed by CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Hwan-Seok Choi, M.D, Ph.D., Principal Investigator — Catholic Medical Center Seoul St. Mary's Hospital; Sae Woong Kim, M.D., Ph.D., Principal Investigator — Catholic Medical Center Seoul St. Mary's Hospital
Locations (9):
- South Korea (9):
  - Inje University Ilsan Paik Hospital, Goyang-si
  - National Health Insurance Service Ilsan Hospital, Goyang-si
  - Pusan National University Hospital, Pusan
  - Catholic Medical Center Seoul St. Mary's Hospital, Seoul
  - Ewha Womans University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Catholic university of Korea Uijeongbu St.Mary's Hospital, Uijeongbu-si